CLINICAL TRIAL: NCT05352061
Title: Addressing Psychosocial Comorbidities in HIV Treatment and Prevention: Phase 2b
Brief Title: Addressing Psychosocial Comorbidities in HIV Treatment and Prevention 2b
Acronym: Synk2b
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Steven Safren, Professor, University of Miami
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20210836; 9K24DA040489 (NIH)
Record Dates: First submitted 2022-04-22; First posted 2022-04-28 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Medication Adherence; Mental Health Issue
Keywords: HIV Medication Adherence; Mental Health
MeSH Terms: conditions — Medication Adherence; Psychological Well-Being | interventions — Syndemic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Cognitive Behavioral Therapy (CBT) for Syndemic and Adherence Factors Group (Experimental): Participants in this group will receive the CBT for Syndemics and Adherence Factors intervention for a total of 14 sessions over 4 months.
  Interventions: Behavioral: CBT for Syndemics and Adherence Factors

INTERVENTIONS:
Behavioral: CBT for Syndemics and Adherence Factors — Each hour-long session is conducted via zoom or in person with a study clinician. Sessions focus on HIV medication adherence, coping with life stressors, and managing other challenging situations (e.g., possible traumatic experiences, drug and alcohol use and sexual behavior) that may affect mental or HIV-related health.

SUMMARY:
The purpose of this study is to learn about ways to better support people living with HIV with their HIV treatment and cope with mental health challenges and/or substance use concerns.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18 years or older
2. HIV positive
3. Evidence of uncontrolled virus (e.g., > 20 copies/ml) within the past 12 months as verified by medical record
4. Group 1: (Men who have sex with men (MSM) who have used stimulants within the past 4 months (approximately 10 participants))OR Group 2: transgender women (approximately 10 participants) OR Group 3: Emerging adults between the ages of 18 and 26 (inclusive; approximately 10 participants)

Exclusion Criteria:

1. Unable to provide informed consent due to severe mental or physical illness, cognitive impairment, or substance intoxication at the time of interview
2. Active untreated, unstable, major mental illness (i.e., untreated psychosis or mania) that would interfere with study participation
3. Opinion of the PI that the participant would be at risk for harm to self or others
4. Currently receiving CBT for a psychiatric disorder, or received a course of CBT in the past year.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Three distinct groups will be recruited: 1) Men who have sex with men who use stimulants, 2) transgender women, 3) emerging adults (ages 18-26 years).
Enrollment: 75 (Estimated)
Dates: Start 2022-08-15 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants who completes the follow up assessment | 8 months
  Feasibility will be reported as the percentage of participants who completes the study follow up assessment.

SECONDARY OUTCOMES:
ART Medication Adherence | Up to 8 months
  Antiretroviral Therapy (ART) adherence will be reported as the percentage of participants who reports taking > 80% of their ART from baseline up to follow up visit.
Percentage of participants with undetectable viral load | Up to 8 months
  As assessed via serum blood samples.
Percentage of participants with improvement in syndemic, behavioral health outcomes | Up to 8 months
  Participants with a 2-point reduction in their Diagnostic Interview for Anxiety, Mood and Obsessive Compulsive Disorder (OCD) Related Neuropsychiatric Disorders (DIAMOND) scores from baseline will be reported as having improvement in behavioral health outcome. DIAMOND has a total score ranging from 1-7 with the higher score indicating greater severity.

CONTACTS AND LOCATIONS:
Overall Officials: Steven A Safren, PhD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No